CLINICAL TRIAL: NCT04746924
Title: A Phase 3, Randomized, Double-Blind Study of Ociperlimab, an Anti-TIGIT Antibody, in Combination With Tislelizumab Compared to Pembrolizumab in Patients With Previously Untreated, PD-L1-Selected, and Locally Advanced, Unresectable, or Metastatic Non-Small Cell Lung Cancer
Brief Title: A Study of Ociperlimab With Tislelizumab Compared to Pembrolizumab in Participants With Untreated Lung Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AdvanTIG-302; BGB-A317-A1217-302 (Other: BeiGene); CTR20211476/CTR20211464 (Other: ChinaDrugTrials); 2020-004985-21 (EudraCT Number)
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Non-small Cell Lung Cancer; NSCLC
Keywords: Locally Advanced; Unresectable; Metastatic; Tislelizumab; BGB-A317; Ociperlimab; BGB-A1217; Pembrolizumab; Anti-TIGIT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — tislelizumab; pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Tislelizumab plus Ociperlimab (Experimental): Participants will receive tislelizumab 200 milligrams (mg) intravenously followed by ociperlimab 900 mg intravenously once every 3 weeks.
  Interventions: Drug: Tislelizumab; Drug: Ociperlimab
- Arm B: Pembrolizumab plus Placebo (Active Comparator): Participants will receive pembrolizumab 200 mg intravenously followed by placebo intravenously once every 3 weeks.
  Interventions: Drug: Pembrolizumab; Drug: Placebo
- Arm C: Tislelizumab plus Placebo (Placebo Comparator): Participants will receive tislelizumab 200 mg intravenously followed by placebo intravenously once every 3 weeks.
  Interventions: Drug: Tislelizumab; Drug: Placebo

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab is a monoclonal antibody formulated for intravenous injection.
  Other Names: BGB-A317
  Arms: Arm A: Tislelizumab plus Ociperlimab; Arm C: Tislelizumab plus Placebo
Drug: Ociperlimab — Ociperlimab is a monoclonal antibody formulated for intravenous injection.
  Other Names: BGB-A1217
  Arms: Arm A: Tislelizumab plus Ociperlimab
Drug: Pembrolizumab — Pembrolizumab is a monoclonal antibody formulated for intravenous injection.
  Other Names: KEYTRUDA
  Arms: Arm B: Pembrolizumab plus Placebo
Drug: Placebo — Placebo infusions will consist of a sterile, normal saline solution.
  Arms: Arm B: Pembrolizumab plus Placebo; Arm C: Tislelizumab plus Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ociperlimab + tislelizumab compared with that of pembrolizumab in adults with PD-L1 high, locally advanced/recurrent or untreated metastatic NSCLC.

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologically or cytologically documented locally advanced or recurrent non-small cell lung cancer (NSCLC) that is not eligible for curative surgery and/or definitive radiotherapy with or without chemoradiotherapy, or metastatic-nonsquamous or squamous NSCLC.
2. No prior systemic treatment for metastatic NSCLC.
3. Agreement to provide archival tissue or fresh biopsy (if archival tissue is not available).
4. Tumors with PD-L1 expressed in ≥ 50% tumor cells.
5. At least 1 measurable lesion as defined per RECIST v1.1.
6. ECOG Performance Status ≤ 1.

Key Exclusion Criteria:

1. Known mutations in the epidermal growth factor receptor (EGFR) gene, anaplastic lymphoma kinase (ALK) fusion oncogene, BRAF V600E, or ROS1.
2. Prior therapy with an anti-programmed cell death protein (anti-PD)-1, anti-PD-ligand (L)-1, anti-PD-ligand-2, anti-T-cell immunoglobulin and ITIM (anti-TIGIT) domain, or any other antibody or drug specifically targeting T-cell costimulation or checkpoint pathways.
3. Active leptomeningeal disease or uncontrolled, untreated brain metastasis.
4. Active autoimmune diseases or history of autoimmune diseases that may relapse.

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 662 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to approximately 58 months
  OS will be defined as the time from the date of randomization to the date of death due to any cause.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) As Assessed By Investigators | Up to approximately 58 months
  PFS will be defined as the time from the date of randomization to the date of the first objectively documented tumor progression per RECIST v1.1, or death, whichever occurs first.
Overall Response Rate (ORR) As Assessed By Investigators | Up to approximately 58 months
  ORR will be defined as the proportion of participants with a documented, confirmed complete response or partial response per RECIST v1.1.
Duration Of Response (DOR) As Assessed By Investigators | Up to approximately 58 months
  DOR will be defined as the time from the first determination of an objective response per RECIST v1.1 until the first documentation of progression or death, whichever occurs first.
Health-related Quality Of Life (HRQoL): European Organization For Research And Treatment Of Cancer Quality Of Life Questionnaire Core 30 (EORTC QLQ-C30) | Within 7 days after permanent treatment discontinuation
  HRQoL will be assessed via patient-reported outcomes (PRO) using the EORTC QLQ-C30.
  The EORTC QLQ-C30 (Version 3) consists of Global health status/QoL (score range from 0=very poor to 7=excellent), 5 functioning scales (physical, role, emotional, cognitive, social), 8 symptom scales (fatigue, nausea/vomiting, pain, dyspnea, insomnia, constipation, diarrhea) and financial difficulties with scores ranging from 1 = "Not at all" to 4 = "Very much". For the global health status/QoL and functioning scales, higher scores indicate better outcomes and for symptom scales, lower scores indicate better outcomes.
HRQoL: EORTC Lung Cancer Module Quality of Life Questionnaire Lung Cancer 13 (QLQ-LC13) HRQoL will be assessed via PRO using the EORTC QLQ-LC13. | Within 7 days after permanent treatment discontinuation
  QLQ-LC13 consists of 10 scales, scores ranging from 1 = "not at all" to 4 = "very much", and 2 questions regarding use of pain medication (yes/no) and if yes, did it help (1 = "not at all" to 4 = "very much"). In symptom scales, lower scores indicate better outcomes.
HRQoL: European Quality of Life-5 Level- 5 Dimension (EQ-5D-5L) Questionnaire | Within 7 days after permanent treatment discontinuation
  HRQoL will be assessed via PRO using the EQ-5D-5L. The EQ-5D-5L comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression, and a visual analog scale (VAS). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The VAS records the respondent's self-rated health on a 0 to 100 scale, with 100 = "the best health you can imagine" and 0 = "'the worst health you can imagine". Lower scores in descriptive dimension indicate better HRQoL and higher VAS scores indicates better health state.
Time To Deterioration (TTD) | Within 7 days after permanent treatment discontinuation
  TTD will be analyzed using PRO scores, and will be defined as worsening scores of ≥10 points from baseline for 2 consecutive assessments or 1 assessment followed by death from any cause.
Number Of Participants Experiencing Adverse Events (AEs) | 90 days (±14) after last dose
  The incidence and severity of AEs will be determined according to National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI CTCAE v5.0).

CONTACTS AND LOCATIONS:
Locations (218):
- United States (9):
  - Providence Medical Foundation St Jude Heritage Healthcare, Fullerton, California
  - Valkyrie Clinical Trials, Los Angeles, California
  - Ocala Oncology Center Pl Dba Florida Cancer Affiliates Ocala, Ocala, Florida
  - Advent Health Cancer Institute, Orlando, Florida
  - Goshen Center For Cancer Care, Goshen, Indiana
  - Baptist Health Lexington, Lexington, Kentucky
  - University Medical Center New Orleans West Jefferson Medical Center, New Orleans, Louisiana
  - Metro Minnesota Community Oncology Research Consortium (Mmcorc), Saint Paul, Minnesota
  - West Penn Hospital, Pittsburgh, Pennsylvania
- Argentina (2):
  - Centro Medical Austral, Buenos Aires
  - Centro Para La Atencion Del Paciente Oncologico (Caipo), San Miguel de Tucumán
- Australia (12):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Northern Cancer Institute, St Leonards, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Pindara Private Hospital, Benowa, Queensland
  - The Prince Charles Hospital, Chermside, Queensland
  - Mater Cancer Care Centre, South Brisbane, Queensland
  - John Flynn Private Hospital, Tugun, Queensland
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - Ballarat Health Services, Ballarat, Victoria
  - Monash Health, Clayton, Victoria
  - Western Health Sunshine Hospital, St Albans, Victoria
  - St John of God, Murdoch, Murdoch, Western Australia
- Brazil (6):
  - Instituto Dor de Pesquisa E Ensino Distrito Federal, Brasília
  - Hospital Evangelico de Cachoeiro de Itapemirim, Cachoeiro de Itapemirim
  - Centro de Pesquisas Oncologicas Cepon, Florianópolis
  - Cancer Institute of Ceara, Fortaleza
  - Cepho Centro de Estudos E Pesquisas de Hematologia E Oncologia, Santo André
  - Fundacao Faculdade Regional de Medicina de Sao Jose Do Rio Preto, São José do Rio Preto
- China (52):
  - Anhui Provincial Hospital, Hefei, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Chao Yang Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing Chest Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Army Military Medical University, Chongqing, Chongqing Municipality
  - Daping Hospital, Third Military Medical University, Chongqing, Chongqing Municipality
  - Chongqing University Three Gorges Central Hospital, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Affiliated Cancer Hospital and Institute of Guangzhou Medical University, Guangzhou, Guangdong
  - Cancer Hospital of Shantou University Medical College, Shantou, Guangdong
  - Shenzhen Peoples Hospital, Shenzhen, Guangdong
  - The Peoples Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - The Tumor Hospital Affiliated to Guangxi Medical University, Nanning, Guangxi
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Changzhou No Peoples Hospital, the Affiliated Hospital of Nanjing Medical University Branch Cheng, Changzhou, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Nanjing Chest Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Soochow University Branch Shizi, Suzhou, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Liaoning Cancer Hospital and Institute, Shenyang, Liaoning
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi
  - The Affiliated Hospital of Qingdao University Branch Laoshan, Qingdao, Shandong
  - Weifang Peoples Hospital, Weifang, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Affiliated Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Sichuan Cancer Hospital and Institute, Chengdu, Sichuan
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Affiliated Hospital of North Sichuan Medical College, Nanchong, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Affiliated Cancer Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang
  - Taizhou Hospital of Zhejiang, Taizhou, Zhejiang
  - The Fourth Affiliated Hospital Zhejiang University School of Medicine, Yiwu, Zhejiang
- France (13):
  - Centre Hospitalier de La Cote Basque Saint Leon Service de Pneumologie, Bayonne
  - Centre de Lutte Contre Le Cancer Institut Bergonie, Bordeaux
  - Hopital de La Croix Rousse, Lyon
  - Hopital Louis Pradel, Lyon
  - Icm Val Daurelle Oncologie Medicale, Montpellier
  - Polyclinique de Gentilly, Nancy
  - Hopital Cochin, Paris
  - Chu Hopital Lyon Sud, PierreBenite
  - Hia Begin, Saint-Mandé
  - Chu de La Reunion, Saint-Pierre
  - Centre de Lutte Contre Le Cancer Institut de Cancerologie de Louest Rene Gauducheau, SaintHerblain
  - Chu Nantes Hopital Nord Laennec, SaintHerblain
  - Chu Tours Hopital Bretonneau Service Pneumologie, Tours
- Georgia (10):
  - High Technology Hospital Medcenter Ltd, Batumi
  - Acad Fridon Todua Medical Center Ltd Research Institute of Clinical Medicine Ltd, Tbilisi
  - Israel Georgian Medical Research Clinic Helsicore Ltd, Tbilisi
  - Jsc German Hospital, Tbilisi
  - Institute of Clinical Oncology Ltd, Tbilisi
  - Jsc Evex Hospitals Tbilisi, Tbilisi
  - Tim Tbilisi Institute of Medicine Ltd, Tbilisi
  - Caucasus Medical Centre Ltd, Tbilisi
  - Multiprofile Clinic Consilium Medulla Ltd, Tbilisi
  - Oncology Research Center Ltd, Tbilisi
- Germany (8):
  - Universitaetsklinikum Aachen, Aachen
  - Universitatsklinikum Bonn, Bonn
  - Kliniken Der Stadt Koeln Ggmbh, Cologne
  - Uniklinikum Giessen Marburg, Giessen
  - Lungenclinic Grosshansdorf Gmbh, Grohansdorf
  - Ambulantes Krebszentrum Hamburg, Hamburg
  - Munchen Klinik Bogenhausen, Munich
  - Agaplesion Diakonieklinikum Rotenburg Gemeinnutzige Gmbh, Rotenburg (Wümme)
- Italy (3):
  - Azienda Ospedaliera Universitaria Policlinico Santorsola Malpighi, Bologna
  - Azienda Ospedaliera Papardo, Messina
  - Aou San Luigi Gonzaga, Orbassano
- Japan (23):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Hirosaki University Hospital, Hirosaki, Aomori
  - Nho Shikoku Cancer Center, Matsuyama, Ehime
  - Kurume University Hospital, Kurume, Fukuoka
  - National Hospital Organization Shibukawa Medical Center, Shibukawa, Gunma
  - Kobe University Hospital, Kobe, Hyōgo
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Hyogo Medical University Hospital, Nishinomiyashi, Hyōgo
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Miyagi Cancer Center, Natorishi, Miyagi
  - Okayama University Hospital, Okayama, Okayama-ken
  - Kansai Medical University Hospital, Hirakata, Osaka
  - National Hospital Organization Kinki Chuo Chest Medical Center, Sakai, Osaka
  - Kindai University Hospital, Sayama, Osaka
  - Osaka Toneyama Medical Center, Toyonaka, Osaka
  - Jichi Medical University Hospital, Shimonotsuke, Tochigi
  - Dokkyo Medical University Hospital, Shimotsugagun, Tochigi
  - Tochigi Cancer Center, Utsunomiya, Tochigi
  - Nippon Medical School Hospital, Bunkyoku, Tokyo
  - Cancer Institute Hospital of Jfcr, Kotoku, Tokyo
  - Hiroshima University Hospital, Hiroshima
  - Niigata Cancer Center Hospital, Niigata
- Netherlands (5):
  - Meander Medisch Centrum, Amersfoort
  - Rijnstate, Arnhem
  - Ziekenhuis St Jansdal, Harderwijk
  - Stichting Zuyderland Medisch Centrum, Heerlen
  - Isala Klinieken Zwolle, Zwolle
- Poland (6):
  - Uniwersytecki Szpital Kliniczny W Bialymstoku, Bialystok
  - Centrum Terapii Wspoczesnej, Lodz
  - Wielospecjalistyczne Centrum Onkologii I Traumatologii Im M Kopernika W Lodzi, Lodz
  - Wielkopolskie Centrum Pulmonologii I Torakochirurgii, Poznan
  - Przychodnia Med Polonia Sp Z Oo, Poznan
  - Etg Zamosc, Zamość
- Russia (8):
  - Arkhangelsk Regional Clinical Oncological Dispensary, Arkhangelsk, Arkhangelskaya oblast
  - State Autonomous Healthcare Institution Republican Clinical Oncological Dispensary of the Republic, Ufa, Bashkortostan Republic
  - State Budgetary Healthcare Institution Regional Oncology Dispensary Number, Magnitogorsk, Chelyabinsk Oblast
  - Vitamed Llc, Moscow, Moscow
  - State Budgetary Healthcare Institution Nizhny Novgorod Regional Clinical Oncology Dispensary, Nizhny Novgorod, Nizhny Novgorod Oblast
  - Bih of Omsk Region Clinical Oncology Dispensary, Omsk, Omsk Oblast
  - State Budgetary Healthcare Institution Samara Regional Clinical Oncology Dispensary, Samara, Samaraskaya Oblast'
  - Llc Av Medical Group, Saint Petersburg, Sankt-Peterburg
- South Korea (8):
  - Chungbuk National University Hospital, Cheongju-si, Chungcheongbukdo
  - Keimyung University Dongsan Hospital, Dalseogu, Daegu Gwang'yeogsi
  - The Catholic University of Korea Bucheon St Marys Hospital, Bucheon-si, Gyeonggi-do
  - Cha Bundang Medical Center, Cha University, Gyeonggido, Gyeonggi-do
  - The Catholic University of Korea, St Vincents Hospital, Suwon, Gyeonggi-do
  - Kyungpook National University Chilgok Hospital, Daegu, Gyeongsangbukdo
  - The Catholic University of Korea, Eunpyeong St Marys Hospital, Eunpyeonggu, Seoul Teugbyeolsi
  - Severance Hospital Yonsei University Health System, Seoul, Seoul Teugbyeolsi
- Spain (24):
  - Hospital Universitario Fundacion Alcorcon, Alcorcón
  - Hospital Del Mar, Barcelona
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Hospital Universitario Vall Dhebron, Barcelona
  - Hospital Universitari Quiron Dexeus, Barcelona
  - Hospital General Universitario de Elche, Elche
  - Ico Girona, Girona
  - Hospital Universitario de Jaen, Jaén
  - Complejo Hospitalario Universitario Insular Gran Canaria, Las Palmas
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Clinico San Carlos, Madrid
  - Start Madrid Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Doce de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitario Virgen de La Victoria, Málaga
  - Hospital General Universitario Morales Meseguer, Murcia
  - Complexo Hospitalario Universitario de Ourense, Ourense
  - Hospital Universitari Son Espases, Palma de Mallorca
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Universitario Nuestra Senora de Valme, Seville
  - Hospital Arnau de Vilanova, Valencia
  - Hospital Universitari I Politecnic La Fe, Valencia
- Taiwan (7):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei
  - Taipei Tzu Chi Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
  - National Taiwan University Hospital Yunlin Branch, Yunlin
- Thailand (7):
  - Siriraj Hospital, Bangkok
  - Songklanagarind Hospital (Prince of Songkhla University), Hat Yai
  - Chulabhorn Research Institute, Lak Si
  - Srinagarind Hospital (Khon Kaen University), Muang
  - Maharaj Nakorn Chiang Mai Hospital (Chiang Mai University), Muang
  - Phramongkutklao Hospital, Ratchathewi
  - Rajavithi Hospital, Ratchathewi
- Turkey (Türkiye) (12):
  - Acibadem Adana Hospital, Adana
  - Baskent University Practice and Research Hospital Adana Medical Oncology Department, Adana
  - Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital, Ankara
  - Memorial Ankara Hospital, Ankara
  - Inonu Universitesi Tip Fakultesi, Battalgazi
  - Tr Trakya University Health Research and Application Center (Hospital), Edirne
  - Iu C, Clinical Research Excellence Application and Research Center, Istanbul
  - Tr Ministry of Health Goztepe Prof Dr Suleyman Yalcin City Hospital, Istanbul
  - Ege University Medical Faculty, Izmir
  - Kocaeli Universitesi Tip Fakultesi, Kocaeli
  - Necmettin Erbakan University Selcuklu Faculty of Medicine, Meram
  - Mersin City Hospital, Mersin City Hospital
- Ukraine (3):
  - Medical Center of Limited Liability Company Mriya Med Service, Kryvyi Rih
  - Communal Non Profit Enterprisecentral Municipal Clinical Hospital of Uzhhorod City Council, Uzhhorod
  - Zakarpatska Regional Clinical Oncological Center, Uzhhorod

IPD SHARING:
Plan to Share IPD: Yes